CLINICAL TRIAL: NCT03259958
Title: A Study to Assess the Steady-State Bioequivalence of Once-Weekly Corplex™ 10mg Donepezil Transdermal Delivery System Compared to Daily Oral Administration of Aricept®
Brief Title: A Bioequivalence Study of Corplex™ Donepezil Transdermal Delivery System Compared to Aricept®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-16010
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donepezil TDS (Experimental): Corplex Donepezil TDS 5 mg/day followed by Donepezil TDS 10mg/day applied weekly for 5 consecutive weeks
  Interventions: Drug: Donepezil TDS
- Aricept (Active Comparator): Aricept 5 mg/day followed by Aricept 10 mg/day once daily for 5 consecutive weeks
  Interventions: Drug: Aricept

INTERVENTIONS:
Drug: Donepezil TDS — Donepezil Hydrochloride Transdermal Delivery System
  Arms: Donepezil TDS
Drug: Aricept — Aricept Tablet
  Arms: Aricept

SUMMARY:
A study to assess the steady-state bioequivalence of once-weekly Corplex™ Donepezil 10 mg Transdermal Delivery System (TDS) compared to daily administration of Aricept®

DETAILED DESCRIPTION:
Open label, randomized, 2-period, multiple-dose crossover study.

Approximately 86 healthy, adult male and female subjects will be enrolled.

Subjects will be randomized to 1 of 2 treatment sequences prior to the first study product treatment in treatment period 1.

For each treatment period; subjects will receive donepezil for 5 consecutive weeks. Blood samples for donepezil PK will be collected pre-dose through week 10.

Adhesion and skin irritation will be monitored throughout TDS treatments. Safety will be monitored throughout the study by adverse event reporting, repeated clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female
* Body mass index ≥ 18.0 and ≤ 32.0 kg/m2 at screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the Investigator
* Have a Fitzpatrick skin type of I, II or III or have skin colorimeter scores equivalent to the allowed Fitzpatrick skin type

Key Exclusion Criteria:

* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds (including piperidine derivatives and other cholinesterase inhibitors)
* Has intolerance to venipuncture and/or inability to comply with the extensive blood sampling required for this study or does not have suitable veins in both arms
* Potential for occupational exposure to anticholinesterase agents.
* Female subjects with a positive pregnancy test or lactating
* Positive urine drug or alcohol results
* Estimated creatinine clearance in non-elderly subjects <80 mL/min at screening and in elderly subjects (i.e., ≥55 years of age) <60 mL/min at screening
* Hemoglobin value of less than 11.5 g/dl for females, 13.0 g/dl for males at screening and first check-in
* Any of the following drugs for 28 days prior to the first dose of study drug in Treatment Period 1 and throughout the study:

  * significant inducers of cytochrome P450 (CYP) enzymes and/or P-glycoprotein;
  * anti-inflammatory drugs or cyclooxygenase 2 (COX-2) analgesic;
  * beta-blockers;
  * anti-fungal medications;
  * anti-histamines;
  * cholinergics and anti-cholinergics;
  * oral corticosteroids;
  * Prolia;
  * adjuvant analgesics
* Muscle relaxants, anti-Parkinsonian or neuroleptic medications prior to the first dose of study drug
* History or presence of excessive hairy skin on application sites as deemed by the Investigator to potentially interfere with drug absorption
* History or presence of significant skin damage, diffuse skin diseases, scars, tattoos on the application sites or other skin disturbances as deemed by the Investigator to potentially interfere with drug absorption or irritation assessments
* Use of donepezil hydrochloride or related drugs within 30 days prior to the first study drug administration
* Participation in another clinical study within 30 days prior to the first study drug administration
* Clinically significant depression symptoms or suicidal ideation or behavior as determined by the Investigator

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
PK, AUC | Blood samples for donepezil PK will be collected pre dose until the end of each treatment period, approximately 10 weeks total
  To assess the plasma concentration (AUC) of once-weekly Corplex Donepezil (TDS) compared to once-daily (QD) administration of Aricept (donepezil hydrochloride [HCl]).
PK, Cmax | Blood samples for donepezil PK will be collected pre dose until the end of each treatment period, approximately 10 weeks total
  To assess the maximum observed concentrations (Cmax) of once-weekly Corplex Donepezil (TDS) compared to once-daily (QD) administration of Aricept (donepezil hydrochloride [HCl]).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Daily during 5 week treatment period and during the 5 week follow-on period
  General Safety (AE and SAE as reported by subject following guidance CTCAE v4.0)
PI assessment of local skin irritation response to TDS | 0.5hr, 24hr, 48hr and 72hr after each TDS removal. (5 consecutive weeks)
  To evaluate the safety and tolerability (including local skin irritation) of once-weekly Corplex Donepezil TDS. Dermal Response assessed using 8 point categorical scale. Other effects assessed using a 6 point scale.
PI assessment of TDS Adhesion | Daily during 5 week treatment period
  Adhesion data will be collected during each 7-day patch wear period throughout 5 week treatment period. Percent adherence will be assessed using 12 point categorical scale.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion
Locations (1):
- Celerion Inc., Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No Plans